CLINICAL TRIAL: NCT02712749
Title: Use of Binaural Beat Premedication Reduces Post-operative Morphine Consumption in Elderly Patient Submitted to Knee Surgery
Brief Title: Use of Binaural Beat Premedication in Elderly Submitted to Major Orthopedic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Toscana Nord Ovest (Other)
Responsible Party: Principal Investigator, Alessandro Tani, Medical Doctor, Azienda USL Toscana Nord Ovest
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IDE
Record Dates: First submitted 2016-03-04; First posted 2016-03-18 (Estimated); Last update posted 2019-04-01 (Actual); Status verified 2018-03

CONDITIONS: Anxiety; Postoperative Pain; Morphine Consumption
Keywords: Binaural Beat; Elderly; preoperative medication; postoperative merphine consumption; postoperative pain
MeSH Terms: conditions — Anxiety Disorders; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A : Sound with Binaural Beats (Experimental): Acoustic frequencies of 256 Hz in one ear and 260 Hz in the opposite ear producing a binaural beat of 4 Hz through generated by the software "Gnaural" in stereo option
  Interventions: Device: Sound with Binaural Beats
- Group B : Sound without Binaural Beats (Active Comparator): Acoustic frequencies of 256 Hz in both ears to perceive one tone without beats generated by the software "Gnaural" in mono option
  Interventions: Device: Sound without Binaural Beats

INTERVENTIONS:
Device: Sound with Binaural Beats — Acoustic frequencies of 256 Hz in one ear and 260 Hz in the opposite ear producing a binaural beat of 4 Hz generated by the special program Gnaural in stereo option
  Arms: Group A : Sound with Binaural Beats
Device: Sound without Binaural Beats — Acoustic frequencies of 256 Hz in both ears to perceive one tone without beats generated by the program Gnaural in mono option
  Arms: Group B : Sound without Binaural Beats

SUMMARY:
The Investigators verify the effectiveness of "Binaural Beats" as premedication instrument in elderly patients submitted to orthopedic surgery to reduce anxiety , post operative pain and morphine consumption

DETAILED DESCRIPTION:
Need for surgery is increasing among elderly population, for increase in average life expectancy and for improved in surgical and anesthetic techniques.

A big problem in this kind of patients is the high incidence of delirium and cognitive impairment in post-operative period , which increase with age, depending on the type of intervention (especially Orthopaedics and Cardiac Surgery) and the administration of some agents, particularly sedatives and opioids .

Premedication is usually carried using anxiolytic and / or narcotic drugs in order to reduce anxiety and discomfort related to the intervention and anesthesia. The preoperative anxiety in fact increases the demand for intra and post operative anesthetics and analgesics and contribute to increase the post operative pain. For this reason the use of a pharmacological premedication is controversial in elderly patient, for the risk of side effects of drugs on one side, and for the other to the discomfort resulting from the increased level of anxiety in absence of premedication. .

Some recent surgical guidelines warn against premedication drug in patients over sixty-five, considering that occurrence of delirium and cognitive impairment may worsen the prognosis, limiting the use of such drugs to what is strictly necessary and only in the immediacy of the surgical act.

To reduce perioperative pain and anxiety , some authors used "Binaural Beats". This simple technique , described for the first time since by Gerald Oster , include the presentation of two acoustic stimuli with similar frequencies through the two channels of stereo headphones. The interference of their waves which occurs at the level of the central nervous system, produces a composite signal with a frequency resulting from the difference of the two original frequencies. For example if you give an acoustic stimulus of 100 Hz to an ear and simultaneously administering another acoustic stimulation of 104 Hz to the opposite ,ear the person who listens to these stimuli will perceive a "Binaural Beat" of 4 Hz caused by the difference between the two frequencies. These Binaural Beats are of interest because they have been thought to cause hemispheric synchronization and influence the EEG frequency like light stimulation .

Binaural Beats have already been used in humans undergoing outpatient surgery in uro-gynecological and have been shown to help increase patient comfort by reducing the state of anxiety and pain without interfering negatively with postoperative functional recovery .

In this study, we applied BBs as premedication in elderly patients who underwent major orthopaedic surgery aimed to reduce anxiety , postoperative pain and morphine consumption.

Feeling/level of anxiety is evaluated using STAI Y1 . This scale is a psychological inventory that consists of 20 questions on a self-report of anxiety about an event.

Feeling/level of pain is evaluated with the use of Numerical Rating Scale (NRS) .It consist to asking the patients to report her/his feeling of pain using an eleven-point scale : 0 = no pain, 10 most severe imaginable pain.

Cumulative morphine consumpion is evaluated through PCA registration. Patient Controlled Analgesia (PCA) is an electronic device that allows a patients to activate intravenous administration of morphine to themselves during the post-operative period. Each request and drug administration is automatically recorded by the device.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 65 years aged candidated to elective major orthopedic surgery
* Stable hemodynamic and clinical conditions (ASA 1/2, Goldman Desky Class 1)
* Absence of cognitive impairment (MMSE greater than 24)
* Valid consent expression to the study participation
* No history of epilepsy and other chronic neurological diseases that may interfere with the study procedures.
* Good collaboration in activities provided by the study
* No abnormalities at audiometric testing for the frequencies between 256 and 260 Hz.

Exclusion Criteria:

* Insufficient level of cooperation or hearing loss
* Contraindications to the use of binaural beats (a history of epilepsy)
* Treatment with anti-anxiety drugs or major tranquillizers
* Clinical Instability defined as the inclusion criteria
* Denial of informed consent to participate in the study
* Presence of cognitive impairment (MMSE less than or equal to 24)
* Presence of neurological diseases or neurological damage that interfere with the study procedures.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-28 (Actual)

PRIMARY OUTCOMES:
Reduction on postoperative morphine consumption | in the first post-operative day
  Difference of cumulative morphine consumption between Binaural Beat group vs Control group through patient-controlled analgesia device (PCA)

SECONDARY OUTCOMES:
Reduction in the level of preoperative anxiety assessed by State Anxiety inventory (STAI-1) | at 20 minutes after a binaural beat listening session
  Measurement of anxiety assessed by STAI-1 after a 20 minutes of binaural beat listening session and comparison between the two groups . The State- Trait Anxiety Inventory is a validated 40-item self-report measure that contains 20 items measuring state anxiety (STAI-1) and 20 items measuring trait anxiety (STAI-2).Scores for state and trait components each range from 20 to 80 with a higher score corresponding to higher anxiety levels.
  The anxiety level is considered low when the STAI is between 20 and 40, moderate between 41 and 60, high between 61 and 80

OTHER OUTCOMES:
Postoperative pain reduction | NRS mesurements at 8, 16 and 24 hours after surgery
  Comparison of the mean value of Numerical Rating Scale (NRS) in three measurements on the first post-operative day between the treated group and control. Numerical Rating Scale (NRS) method consist to asking the patients to report her/his feeling of pain using an eleven-point scale : 0 = no pain, 10 most severe imaginable pain.
  NRS scores ≤ 3 correspond to mild, scores of 4-6 to moderate and scores ≥7 to severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Tani, MD, Principal Investigator — Usl Area Vasta Nord Ovest
Locations (1):
- Santa Maria Maddalena Hospital, Volterra, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deiner S, Silverstein JH. Postoperative delirium and cognitive dysfunction. Br J Anaesth. 2009 Dec;103 Suppl 1(Suppl 1):i41-46. doi: 10.1093/bja/aep291. PMID 20007989
- [Background] Kain ZN, Sevarino F, Alexander GM, Pincus S, Mayes LC. Preoperative anxiety and postoperative pain in women undergoing hysterectomy. A repeated-measures design. J Psychosom Res. 2000 Dec;49(6):417-22. doi: 10.1016/s0022-3999(00)00189-6. PMID 11182434
- [Background] Ozalp G, Sarioglu R, Tuncel G, Aslan K, Kadiogullari N. Preoperative emotional states in patients with breast cancer and postoperative pain. Acta Anaesthesiol Scand. 2003 Jan;47(1):26-9. doi: 10.1034/j.1399-6576.2003.470105.x. PMID 12492793
- [Background] Padmanabhan R, Hildreth AJ, Laws D. A prospective, randomised, controlled study examining binaural beat audio and pre-operative anxiety in patients undergoing general anaesthesia for day case surgery. Anaesthesia. 2005 Sep;60(9):874-7. doi: 10.1111/j.1365-2044.2005.04287.x. PMID 16115248
- [Background] Kliempt P, Ruta D, Ogston S, Landeck A, Martay K. Hemispheric-synchronisation during anaesthesia: a double-blind randomised trial using audiotapes for intra-operative nociception control. Anaesthesia. 1999 Aug;54(8):769-73. doi: 10.1046/j.1365-2044.1999.00958.x. PMID 10460529
- [Background] Dabu-Bondoc S, Vadivelu N, Benson J, Perret D, Kain ZN. Hemispheric synchronized sounds and perioperative analgesic requirements. Anesth Analg. 2010 Jan 1;110(1):208-10. doi: 10.1213/ANE.0b013e3181bea424. Epub 2009 Oct 27. PMID 19861358
- [Background] Goodin P, Ciorciari J, Baker K, Carey AM, Harper M, Kaufman J. A high-density EEG investigation into steady state binaural beat stimulation. PLoS One. 2012;7(4):e34789. doi: 10.1371/journal.pone.0034789. Epub 2012 Apr 9. PMID 22496862
- [Background] Le Scouarnec RP, Poirier RM, Owens JE, Gauthier J, Taylor AG, Foresman PA. Use of binaural beat tapes for treatment of anxiety: a pilot study of tape preference and outcomes. Altern Ther Health Med. 2001 Jan;7(1):58-63. PMID 11191043
- [Background] Schmidt WD, O'Connor PJ, Cochrane JB, Cantwell M. Resting metabolic rate is influenced by anxiety in college men. J Appl Physiol (1985). 1996 Feb;80(2):638-42. doi: 10.1152/jappl.1996.80.2.638. PMID 8929609
- [Background] Millar K, Jelicic M, Bonke B, Asbury AJ. Assessment of preoperative anxiety: comparison of measures in patients awaiting surgery for breast cancer. Br J Anaesth. 1995 Feb;74(2):180-3. doi: 10.1093/bja/74.2.180. PMID 7696068
- [Background] Dolin SJ, Cashman JN, Bland JM. Effectiveness of acute postoperative pain management: I. Evidence from published data. Br J Anaesth. 2002 Sep;89(3):409-23. PMID 12402719
- [Background] Hollenberg SM. Preoperative cardiac risk assessment. Chest. 1999 May;115(5 Suppl):51S-57S. doi: 10.1378/chest.115.suppl_2.51s. PMID 10331334
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- See also: gnaural software generating binaural beat — http://gnaural.sourceforge.net/